CLINICAL TRIAL: NCT06725134
Title: Impact of Therapy Dogs on Anxiety and Behavior of Pediatric Dental Patients During Local Anesthesia: A Randomized Controlled Trial
Brief Title: Impact of Therapy Dogs on Child Anxiety and Behavior During Local Anesthesia for Dental Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, James R. Boynton, Clinical Professor of Dentistry, Department of Pediatric Dentistry, School of Dentistry, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HUM00260476
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Situational Anxiety; Behavior
Keywords: Animal assisted therapy; Pediatric dentistry; Local anesthesia
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Standard-of-care basic behavior guidance during local anesthesia
  Interventions: Behavioral: Standard-of-care basic behavior guidance
- Therapy dog presence (Experimental): Therapy dog present during local anesthesia administration
  Interventions: Behavioral: Therapy dog presence

INTERVENTIONS:
Behavioral: Therapy dog presence — A trained therapy dog will be present during the child's dental appointment. The dog will be in the operatory as the child enters the room and will lie on the child during injection of local anesthesia.
  Arms: Therapy dog presence
Behavioral: Standard-of-care basic behavior guidance — Basic behavior guidance as defined by the American Academy of Pediatric Dentistry includes strategies to help children cope through potentially stressful dental procedures. These strategies include tell-show-do, positive reinforcement, parental presence, and nitrous oxide/oxygen analgesia, among others.
  Arms: Control

SUMMARY:
Therapy dogs in dental offices might help anxious children during dental care. Therapy dogs might help children during injection of local anesthetic, when we inject numbing medication before working on the teeth. The goal of this study is to learn if having a therapy dog with a child during the injection of numbing medication helps children to be more comfortable at the dentist's office. This study is of children who need dental care using local anesthesia. Study participant's behavioral reactions and heart rate during injection of local anesthetic with and without having a therapy dog present will be recorded and children and their guardians will be asked a few short questions about the injection and therapy dog after injection.

DETAILED DESCRIPTION:
Children undergoing dental restorative or surgical procedures require injection of local anesthetic. The injection procedure is often the most anxiety-producing stimulus for children during dental care, when children demonstrate the highest level of emotional distress. Several studies have investigated various interventions, such as distraction, hypnosis, and cognitive behavioral therapy to ease this stress. Animal-assisted therapy (e.g. the presence of a therapy dog) may be a promising strategy for managing anxiety in young dental patients. However, no studies have explored the potential benefits of using therapy dogs specifically during the administration of local anesthesia in pediatric dental patients. The objective of this randomized controlled trial is to investigate the effects of therapy dogs on pediatric dental patients during local anesthesia administration.

ELIGIBILITY:
Inclusion Criteria:

* Age range: children aged 4- to 12-years
* Health status: healthy children without significant medical conditions (ASA I or ASA II)
* Dental procedure: children scheduled for at least two dental procedures requiring local anesthesia
* Consent: written informed consent from the parent or legal guardian
* Verbal assent from potential subjects age 4-9 years; written assent for children age 10-12 years

Exclusion Criteria:

* Allergies: children with known allergies to dogs or animal dander
* Children with a fear or phobia of dogs
* Children with a behavioral disorder which may negatively impact response to the presence of a therapy dog
* Previous exposure: children who have previously undergone dental procedures with local anesthesia in the presence of a therapy dog
* Medical conditions: children with medical conditions that might affect their vital signs independently of the dental procedure (e.g., heart conditions)
* Parental discomfort: cases where parents are uncomfortable with the presence of a therapy dog during the procedure
* Advanced behavior guidance is indicated: children whose behavior for dental examination is classified as "Definitely Negative" (Frankl 1)

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Behavior (Face, Legs, Activity, Cry, and Consolability scale) | Every 30 seconds from entry into the operatory through one-minute following injection of local anesthesia
  The subject's behavior from entry into the operatory through one minute following administration of local anesthesia will be evaluated and recorded using the Face, Legs, Activity, Cry, and Consolability (FLACC) scale, with each category scored from 0 to 2. The higher the total score, which ranges from 0 to 10, indicates more distress.

SECONDARY OUTCOMES:
Heart rate | Every 30 seconds from entry into the operatory through one-minute following injection of local anesthesia
  The subject's heart rate will be monitored and recorded every 30 seconds from entry into the operatory through one minute following administration of local anesthesia.
Anxiety assessment (Modified Faces version of the Modified Child Dental Anxiety scale) | Upon entering the operatory and after administration of local anesthesia
  The subject will be asked to complete an anxiety assessment using the revised modified faces version of the modified child dental anxiety scale (MCDASF). This questionnaire has two questions which are each answered on a five-point scale (range 1-5 for each question for a total range of 2-10). Higher values represent more distress.
Parent questionnaire | Following injection of local anesthetic
  The subject's parent will be asked four questions regarding their child's anxiety and the therapy dog (if present). These four questions are not scaled. The questions are: Do you think your child was anxious for local anesthesia? Y/N; Do you think the therapy dog reduced your child's dental anxiety during local anesthesia? Yes/No; Would you want a therapy dog present for future dental treatment appointments? Yes/No; How do you think your child fees post-local anesthesia? Very Anxious/Anxious/Neutral/Calm/Very Calm.

CONTACTS AND LOCATIONS:
Overall Officials: James R. Boynton, DDS, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Dentistry Children's Clinic, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No